CLINICAL TRIAL: NCT06076109
Title: Early Awake Alterning Prone Positioning Combined With Non-invasive Oxygen Therapy in Patients With COVID-19 (APPearl).
Brief Title: Early Awake Alterning Prone Positioning Combined With Non-invasive Oxygen Therapy in Patients With COVID-19.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We do not have more subjects to enter into the study.
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Thierry Hernández Gilsoul, Head of department, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Appearl
Record Dates: First submitted 2023-10-09; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRONE POSITION (Active Comparator): Patients who require supplemental oxygen through a non-invasive device (nasal cannulas or reservoir mask) in the prone position.
  Interventions: Other: Prone position
- STANDARD TREATMENT (Placebo Comparator): Patients who require supplemental oxygen through a non-invasive device (nasal cannulas or reservoir mask) in the supine position with the head of the bed between 30-60º.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Prone position — Patients who require supplemental oxygen through a non-invasive device (nasal cannulas or reservoir mask) in the prone position.
  Arms: PRONE POSITION
Other: Standard treatment — Patients who require supplemental oxygen through a non-invasive device (nasal cannulas or reservoir mask) in the supine position with the head of the bed between 30-60º.
  Arms: STANDARD TREATMENT

SUMMARY:
Introduction: The disease caused by the new coronavirus (COVID-19) represents a pandemic with significant affectation in our country, generating critical illness in around 5% of the patients who present this disease at an international level, with the requirement of invasive mechanical ventilation being the main cause of admission to intensive care units (UTI).

Objective: to evaluate the utility of using the prone position in patients with hypoxemic respiratory failure with COVID-19 who are with non-invasive oxygenation devices to reduce the need for invasive mechanical ventilation and mortality in this population.

Material and methods: a controlled and randomized clinical trial will be carried out, which will include patients who come to the institution for medical attention with a confirmed or suspected diagnosis of COVID-19 with a severe presentation, hypoxemic respiratory failure, and non-existent oxygen therapy. invasive with a FiO2 contribution ≥40%. The patients enter 2 follow-up groups: an intervention group in which the prone position maneuver performed by the patient himself will be implemented, and another group where the patients will remain supine with the head of their bed between 30-60º. The demographic and clinical variables of these patients will be described. The primary outcome to be evaluated will be the proportion of patients requiring orotracheal intubation during their hospital stay. The secondary outcomes that will be evaluated will be hospital mortality, development of ARDS, and changes in oxygenation by determining SpO2 and SpO2/FiO2 on admission and at 1, 6, 12, 24, 48, and 72 hours after inclusion in the protocol. , as well as PaO2/FiO2 on admission and at 24 hours; the time interval between inclusion in the protocol and orotracheal intubation, use of non-invasive ventilatory therapies, days of hospital stay, days of stay in intensive care, days free of mechanical ventilation, development of acute organ failure during hospitalization and complications related to the treatment with the prone position.

ELIGIBILITY:
Inclusion Criteria:

* - Age greater than or equal to 18 years at the time of the initial evaluation.
* Patient hospitalized in non-critical areas, with at least 12 hours and no more than 48 hours of hospital stay at the time of randomization with a clinical picture of severe COVID-19, according to the following:

  o Patient with symptoms of COVID-19, who meets ≥1 of the following criteria:
  * Tachypnea (≥30 breaths per minute)
  * Arterial oxygen saturation (SaO2) in ambient air (FiO2 21%) less than or equal to 93% at sea level (89% in Mexico City), with supplemental oxygen requirements ≥4 liters per minute.
  * Arterial pressure ratio of Oxygen and Fraction of Inspired Oxygen (PaFi) <300
  * Pulmonary infiltrates in imaging study covering >50% of lung fields, within the last 24 to 48 hours.
  * Administration of supplemental oxygen through a device that provides FiO2 ≥40% (nasal cannulas at a flow of 5 liters or reservoir mask
* The participant understands and agrees with the intervention, randomization and follow-up that will be given during hospitalization and after discharge home and signs the informed consent document prior to randomization

Exclusion Criteria:

* The patient does not wish to participate in the study

  * Patients in palliative care
  * Patients with an indication for orotracheal intubation defined by the presence of at least 2 of the following criteria:

    * Refractory hypoxemia (SaO2 <90% or PaO2 ≤60% with an oxygenation device providing FiO2 ≥60%) for ≥5 minutes without technical failure of the monitoring or oxygenation device
    * Respiratory rate ≥35 breaths per minute
    * Persistent clinical signs of respiratory fatigue: use of accessory muscles of respiration and thoraco-abdominal dissociation
    * acute respiratory acidosis (PH ≤ 7.25, PaCO2 >45 mmHg)
    * abundant respiratory secretions with inability for adequate expectoration by the patient or OR indication for orotracheal intubation due to the presence of 1 of the following criteria:
    * Airway protection requirement: acute altered mental status (ECG <10 points) with absence of airway protection reflexes, active hemoptysis or hematemesis, or airway obstruction. Patients with hypoxemic respiratory failure presenting state unresolved shock (need for resuscitation with intravenous fluids and/or requirement for administration of vasopressors), and unstable arrhythmias (bradycardia or tachycardia)
  * Patients with unresolved shock (resuscitation phase or norepinephrine dose ≥0.15 mcg/kg/min), and unstable arrhythmias (bradycardia or tachycardia).
  * Agitation or acute alteration of the mental state (ECG <10 points) that do not allow the cooperation of the patient for his mobilization to the prone position
  * Instability of the pelvis, spine, or femur from recent surgery or trauma
  * Anatomical alterations that limit the adoption of the prone position (severe xiphoscoliosis, contractures in the extremities, other alterations).
  * Abdominal surgery in the last 15 days
  * Chest injury or chest surgery in the last 15 days or Pregnancy or intracranial hypertension
  * Deep vein thrombosis in the last 2 days
  * Cardiac pacemaker placement in the last 2 days
  * Chest tube with air leak or recent facial trauma or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Orotracheal intubation and invasive mechanical ventilation at 28 days. | 28 days
  The proportion of patients requiring orotracheal intubation and invasive mechanical ventilation at 28 days post-randomization, as well as the proportion of patients who die within this post-randomization time interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico